CLINICAL TRIAL: NCT02553655
Title: Does Remote Ischemic Limb Preconditioning Improve Cerebral Vasomotor Reactivity in Healthy Volunteers?
Brief Title: Remote Ischemic Limb Preconditioning In Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sebastian Koch, Professor of Clinical Neurology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20150648
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Cerebrovascular Disease; Stroke
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4x 5min Limb Preconditioning (Active Comparator): Either the right or left leg of the participant(s) will be made transiently ischemic for 5 minutes following by 5 minutes of rest. This will be repeated for 4 times.
  Interventions: Procedure: 4x 5min Limb Preconditioning
- 3x 10min Limb Preconditioning (Active Comparator): Either the right or left leg of the participant(s) will be made transiently ischemic for 10 minutes following by 5 minutes of rest. This will be repeated for 3 times.
  Interventions: Procedure: 3x 10min Limb Preconditioning
- 3x 10min Sham Preconditioning (Sham Comparator): Either the right or left leg of the participant(s) will be squeezed without causing ischemia for 10 minutes following by 5 minutes of rest. This will be repeated for 3 times.
  Interventions: Procedure: 3x 10min Sham Preconditioning

INTERVENTIONS:
Procedure: 4x 5min Limb Preconditioning — A blood pressure cuff is placed over the upper thigh of the participant(s) and inflated to 30 millimeters of mercury (mmHg) above systolic blood pressure. The loss of pedal pulses is confirmed by palpation. The cuff remains inflated for 5min and is followed by 5 minutes of reperfusion/rest. This will be repeated 4 times.
  Arms: 4x 5min Limb Preconditioning
Procedure: 3x 10min Limb Preconditioning — A blood pressure cuff is placed over the upper thigh of the participant(s) and inflated to 30 mmHg above systolic blood pressure. The loss of pedal pulses is confirmed by palpation. The cuff remains inflated for 10min and is followed by 5 minutes of reperfusion/rest. This will be repeated 3 times.
  Arms: 3x 10min Limb Preconditioning
Procedure: 3x 10min Sham Preconditioning — A blood pressure cuff is placed over the upper thigh of the participant(s) and inflated to 40 mmHg, sufficient to apply pressure but not affect blood flow. The presence of pedal pulses is confirmed by palpation. The cuff remains inflated for 10min and is followed by 5 minutes of rest. This will be repeated 3 times.
  Arms: 3x 10min Sham Preconditioning

SUMMARY:
The investigators would like to determine if remote ischemic leg preconditioning in healthy volunteers improves cerebral vasomotor reactivity as measured by breath holding and transcranial doppler vasomotor reactivity.

DETAILED DESCRIPTION:
This study is to determine if remote ischemic leg preconditioning improves short and long term cerebral vasomotor reactivity in healthy volunteers as measured by breath holding and transcranial doppler vasomotor reactivity. Previous studies on brachial vasomotor reactivity have shown a beneficial effect of remote ischemic preconditioning. It remains uncertain if a similar beneficial effect can be reproduced with cerebral vasomotor testing. Many biological mechanisms and effector pathways triggered by preconditioning have demonstrated endothelial protection and beneficial vascular effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Presence of chronic medical conditions such as diabetes, hypertension, cardiac disease etc.
* Any prescribed medication
* Pregnancy [by history and last menstrual period]
* Any leg injury that would, in the opinion of the investigator, affect preconditioning

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Vasomotor Reactivity to Carbon Dioxide (CO2) | Baseline to 24 hours, Baseline to 48 hours
  Change in vasomotor reactivity to carbon dioxide (CO2) or breath holding from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Koch, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No